CLINICAL TRIAL: NCT04703296
Title: Mindfulness Training in Special Operations Forces (SOF) Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amishi Jha, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201488; W81XWH20C0065 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Change
Keywords: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training (MT) group (Experimental): Receives 4 weeks of mindfulness training followed by a testing session.
  Interventions: Behavioral: MBAT course
- No-training control (NTC) group (No Intervention): Receives 4 weeks of no mindfulness training followed by a testing session.

INTERVENTIONS:
Behavioral: MBAT course — The MBAT will involve:
  (i) 4 weekly 1.5-hour course sessions. The sessions will provide guided exercises, didactic information, and discussions to promote greater mindfulness.
  (ii) Daily mindfulness practice that will be facilitated by the Measuring Mindfulness App (MMA) and/or instructor-delivered mindfulness practices. The daily mindfulness practice will require about 15 minutes to complete.
  Arms: Mindfulness training (MT) group

SUMMARY:
The overarching goal of this study is to develop, deliver, and investigate the utility and feasibility of train-the-trainer delivery of mindfulness training (MT) in support of improved readiness (across cognitive, affective, and social domains of the human dimension) and improve retention of candidates in the SOF qualification pipeline at the U.S. Army John F. Kennedy Special Warfare Center and School (referred to as SWCS).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are between 18 and 65 years of age.
* Individuals who are fluent English speakers.
* Individuals who are active-duty service members.
* Men and women of all races and ethnicities.
* Individuals who are willing and able to consent to participate in the study.
* Individuals who are attending Special Warfare Center and School (SWCS).

Exclusion Criteria:

* Individuals who have a medical or neurological condition that might interfere with performance on the task in the study (e.g., epilepsy)
* Individuals with a history of hospitalization for psychological/mental health issues within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Attentional Performance | Baseline (week 1) to week 6 (after 4-week training interval)
  Attentional Performance as measured by the Sustained Attention Response Task (SART). SART has a range of scores from 0 to 1 with a higher score indicating better accuracy of completing the task.
Change in Working Memory Performance | Baseline (week 1) to week 6 (after 4-week training interval)
  Working Memory Performance as measured by the Working Memory Task with Affective Distracters (WMDA). WMDA has a range of scores from 0 to 100%, with higher scores indicating better accuracy on the task.
Change in Cognitive Failures | Baseline (week 1) to week 6 (after 4-week training interval)
  Cognitive Failures will be measured by the Cognitive Failures Questionnaire (CFQ). CFQ has total score ranging from 0 to 100, with a higher score indicating more cognitive failures.

SECONDARY OUTCOMES:
Change in Positive Affect | Baseline (week 1) to week 6 (after 4-week training interval)
  Positive Affect will be measured by the Positive and Negative Affect Schedule (PANAS-10). The PANAS Positive has a range of scores from 5 to 25, with higher score indicating higher positive mood.
Change in Negative Affect | Baseline (week 1) to week 6 (after 4-week training interval)
  Negative Affect will be measured by the Positive and Negative Affect Schedule (PANAS-10). The PANAS Negative has a range of scores from 5 to 25, with higher score indicating higher negative mood.
Change in Perceived Stress | Baseline (week 1) to week 6 (after 4-week training interval)
  The short version of the Perceived Stress Scale (PSS) will be used assess perceived stress. The 4-item PSS has a range of scores from 0 to 16, with higher score indicating higher level of perceived stress.
Change in Psychological Health | Baseline (week 1) to week 6 (after 4-week training interval)
  Patient Health Questionnaire (PHQ-4) will be used to assess depression and anxiety. PHQ-4 has a range of scores from 0 to 12, with higher scores indicating higher level of depression and anxiety.
Change in Decentering | Baseline (week 1) to week 6 (after 4-week training interval)
  EQ Decentering is an 11-item sub-scale measuring various thoughts and experiences, and the tendency to distance from those. The decentering score ranges from 1 to 55, with a higher score indicating high level of decentering.
Change in Mind Wandering | Baseline (week 1) to week 6 (after 4-week training interval)
  Four Factor Mind Wandering (4FMW) Questionnaire is a 16-item scale that asks participants to indicate how often they experience a situation described in the form of a statement on a 5-point Likert-type scale from never (1) to always (5). 4FMW has a range of scores from 16 to 80, with higher scores indicating greater mind wandering.

OTHER OUTCOMES:
Change in Post-Traumatic Stress Disorder (PTSD) symptomatology | Baseline to week 6 and week 11.
  Post-traumatic Stress Disorder Checklist for military populations (PCL-M) will be used to measure symptoms of PTSD. PCL-M has a range of scores from 17 to 85, with higher scores indicating more PTSD symptoms.
Change in Perspective Taking | Baseline (week 1) to week 6 (after 4-week training interval)
  The Perspective Taking (PT) Subscale from the Interpersonal Reactivity Index (IRI) will be used to assess perspective-taking. The PT Subscale score ranges from 0 to 28, with a higher score indicating greater perspective-taking.
Applied Mindfulness Process Scale | post training at at week 6
  Applied Mindfulness Process Scale measures how often people apply mindfulness practice in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi Jha, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No